CLINICAL TRIAL: NCT01667705
Title: Patient Experience in the CT Scan Suite
Brief Title: To Examine the Effect of a View of Nature on Patient's Stress and Anxiety
Acronym: Skyceiling
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Technical University of Twente (Other)
Responsible Party: Principal Investigator, Trialbureau radiology, Coordinating investigator, Erasmus Medical Center
Other Study IDs: EMCSkyceiling01032012
Record Dates: First submitted 2012-03-01; First posted 2012-08-17 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Stress; Anxiety
Keywords: Stress; Anxiety; Skyceiling; Nature
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SkyCeiling during CT-Suite visit: Patients in the trial group are exposed to the SkyCeiling during their procedure.
- No SkyCeiling during CT-Suite visit: Patients in the trial group are not exposed to the SkyCeiling during their procedure.

SUMMARY:
* Rationale: Recently, research that demonstrates a clear relationship between the built healthcare environment and the health and wellbeing of patients has come available. Patients in a CT scan suite are usually anxious. The environment has been shown to lower stress; a painting or piece of art for example, can capture and hold attention and thereby lower negative thoughts and evoke positive emotions. Sights of nature have demonstrated to be especially effective in recuperating from stress, presumably because the human brain has evolved in a natural environment. The current study will investigate the effects of exposure to nature in the CT scan suite. A SkyCeiling, a large, slightly illuminated, photographic illusion of a real sky view is placed above the CT scan. The main hypothesis of this study is that a sky view will lead to a lower level of anxiety in the CT scan suite.
* Objective: The primary objective of this study is to examine the effect of a view of nature on a patient's stress and anxiety. Secondary objectives are to study the effects of a view of nature on a patient's environmental appraisals of the CT suite, satisfaction with the provided service, and trust in the healthcare provider.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE

   The importance and the potential benefits of well-designed healthcare facilities have been widely acknowledged and recent research clearly demonstrates the relationship between the built healthcare environment and patients' health and well-being (Dijkstra, 2009).

   Encounters with healthcare situations are generally characterized by fear, anxiety, stress, and uncertainty (Mitchell, 2003; Pearson, Maddern, & Fitridge, 2005). Looking at most environments in which these encounters take place, one might rightfully ask how well these healthcare environments satisfy the psychological needs of patients.

   In order to create more beneficial environments, environmental stimuli can be added to (or removed from) the environment to influence the patient in a positive manner. The environment may elicit positive feelings, hold attention and interest, and block or reduce negative thoughts, for example, by the presence of art or a view from a window (R. S. Ulrich, 1984). The purpose of the present study is to improve patients' well-being by adding positive elements to existing healthcare environments, such as pictures of nature.

   Stress is an important factor in healthcare situations and stress reactions can be considered a clinical problem since they often result in negative or worsened medical outcomes (Malkin, 2008). Previous studies (Volicer & Volicer, 1978), for example, found that hospital stress was correlated with changes in heart rate and blood pressure. Other studies showed that psychological stress impairs wound healing in patients (Christian, Graham, Padgett, Glaser, & Kiecolt-Glaser, 2006; Kiecolt-Glaser, Marucha, Malarkey, Mercado, & Glaser, 1995). Elbrecht and colleagues (Elbrecht et al., 2004) studied the effects of perceived stress and cortisol levels on wound healing and demonstrated a considerable negative effect of stress.

   Rabin (2004 in Malkin 2008; personal communication 2008) proposed that pleasant healthcare environments are those that are perceived by the brain as calming, meaning that the stress reactive areas of the brain decrease their activity with a resultant decrease in the concentration of cortisol and norepinephrine in the blood. This results in patients experiencing less pain, having more restful sleep, less anger, less muscle tension, and a lower risk of stroke. Furthermore, Kaplan and Kaplan (R. Kaplan & Kaplan, 1989) state that "the nervous system seems to be structured in such a way that pleasure and pain tend to inhibit each other". A more pleasant healthcare environment could, therefore, result in less stress and anxiety in patients and this should lead to better health and increased feelings of well-being. When speaking about a more pleasant healthcare environment, a wide variety of environmental characteristics come to mind. Variables such as indoor plants and music could help create environments that generate positive feelings and, as a consequence, reduce negative outcomes.

   Nonpharmacological anti-anxiety interventions The advantage of using environmental interventions to lower anxiety is that these kind of interventions do not carry any risk and are not time consuming. Several studies have examined various methods of anxiety reduction in healthcare environments. For example, research has demonstrated the beneficial effects of scents on anxiety and mood in dental patients (Lehrner, Eckersberger, Walla, Poetsch, & Deecke, 2000; Lehrner, Marwinski, Lehr, Johren, & Deecke, 2005) Furthermore, music therapy has successfully been applied to reduce pain and anxiety in patients undergoing various medical procedures, such as children with cancer undergoing lumbar puncture (Thanh Nhan, Nilsson, Hellström, & Bengtson, 2010) and women during caesarian delivery (Chang & Chen, 2005). Sunlight appeared to have beneficial effects on perceived stress (Walch et al., 2005). A recent study (Park & Mattson, 2009) demonstrated that indoor plants in a hospital room can have therapeutic value and serve as a noninvasive and effective complementary medicine for surgical patients. Esthetic enhancements can thus provide unobtrusive and inexpensive stress and anxiety management methods. In this study we propose nature as an anti-anxiety intervention, which possibly has an even stronger effect on anxiety then scent, daylight or music.

   Nature interventions Research on restorative environments suggests that certain environments are capable of promoting recovery from stress. Especially natural settings have these restorative effects (Hartig, Book, Garvill, Olsson, & Garling, 1996). Considering the potential healing properties of nature (Lohr & Pearson-Mims, 2000; R. S. Ulrich, 1984), exposing patients to natural elements may be an effective way of reducing stress. A recent review concluded that viewing nature scenes may decrease pain perceptions by eliciting positive emotional responses and decreasing stress (Malenbaum, Keefe, Williams, Ulrich, & Somers, 2008).

   Ulrich et al. (R. Ulrich et al., 1991) studied the effects of exposure to nature on stress recovery. Participants watched a videotape that induced feelings of stress, and were afterwards exposed to a tape with either a natural or an urban environment. Results demonstrated that individuals recover sooner from stress when exposed to the former (natural) than the latter (urban). Lohr and Pearson-Mims (2000) studied whether the presence of indoor plants would increase pain tolerance. Participants were either placed in a room with plants, a room with non-plant objects (as visually distractive as the plants), or a control room (no objects). Results showed that a significantly larger proportion of respondents in the room with plants were able to keep their hand in the ice water for 5 minutes as compared to the other conditions, suggesting increased pain tolerance by exposure to indoor plants. They also showed that the room with plants was rated more positively (e.g., cheerful, calming, pleasant) than either of the control rooms. The results of these studies support the idea that nature may have beneficial effects on the health and well-being of people.

   Natural elements in the built environment have clearly shown stress-reducing properties, but it is still unclear which underlying mechanism causes this stress-reduction. A potential explanation lies in the theories by Kaplan (S. Kaplan, 1987) and Ulrich (R. S. Ulrich, 1983), which state that people have a tendency to prefer natural settings to built environments. Although these two theories have some important differences (see Hartig et al. (1996) for a discussion), both are based on the same evolutionary assumptions. The preferences for natural settings are assumed to have an evolutionary base; people are to some extent biologically adapted to natural as opposed to built environments. Secondly, it might be argued that nature may be processed more easily and efficiently because the brain and sensory systems evolved in natural environments (Wohlwill, 1983). As a result, humans have an innate tendency to pay attention and respond positively to natural elements (Ulrich et al., 1991). This predisposition to prefer natural elements to man-made objects may be the explanation of the stress-reducing effects of nature. It might thus be hypothesized that natural elements affect feelings of stress through the perceived attractiveness of an environment.

   In a laboratory experiment, Dijkstra et al. (Dijkstra, Pieterse, & Pruyn, 2008) tested this hypothesis and demonstrated the stress-reducing properties of indoor plants in a simulated hospital room. Moreover, this effect was mediated by the perceived attractiveness of the hospital room. The presence of indoor plants in a hospital resulted in participants perceiving the room as more attractive, which in turn resulted in less perceived stress. Considering the potential infection risks of real plants, Dijkstra (Dijkstra, 2009) conducted a second experiment in a figurative painting of a tree was added to a patient room. This second experiment re-confirmed the stress-reducing properties of nature, and replicated the mediating effect of perceived attractiveness on stress. Furthermore, stress is not only reduced by indoor plants, but by a painting of nature as well. An association task revealed that, next to indoor plants, a painting of a tree also activated the concept of nature. This suggests that a mere association with nature could potentially lead to beneficial effects.

   Taken together, nature interventions have shown to be beneficial in a variety of settings. This includes both real and simulated nature interventions. Applying such nature interventions in the CT scan suite might thus lead to beneficial effects in patients.
2. OBJECTIVES

This research project aims to gain insight in how the physical environment of the CT scan suite affects patients' health and well-being. Patients undergoing procedures in a CT scan suite are often anxious and frightened. Stress reactions can be considered a clinical problem since they often result in negative or worsened medical outcomes. Reduction in state anxiety may help to promote relaxation, which in turn is beneficial for a patient's sense of well-being.

Primary Objective: to determine whether a skyceiling lowers stress and anxiety during diagnostic procedures in a CT scan suite.

Secondary Objective(s): to determine whether a skyceiling improves environmental appraisals, mood, satisfaction with the provided service, time perception, and trust in the healthcare provider.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* Able to read and write Dutch
* Able to observe the visual stimuli applied to the ceiling, i.e. normal vision or corrected to normal vision.

Exclusion Criteria:

* Patients who have undergone a CT scan after the SkyCeiling was installed (this is a rare event) are excluded. This because of the fact that these patients might remember the look of the CT unit either with or without the SkyCeiling and could thus become more aware of the intended anxiety-reducing effect of the intervention, or the lack thereof if randomized to the control group.
* Patients who undergo a second scan during the run time of this study (this will be a rare event) will not be included a second time. The data of their first scan remain included.
* Patients who lie with their face down or are otherwise incapable of looking at the ceiling will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 Out-patients, age 18-85, who are scheduled to undergo a thorax and/or abdomen CT scan with intravenous contrast.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
stress and anxiety measured with questionnaires and physiological parameters | 30 minutes During CT-scan visit

SECONDARY OUTCOMES:
environmental appraisals, mood, satisfaction with the provided service, time perception, and trust in the healthcare provider. | 30 minutes during CT-scan visit

CONTACTS AND LOCATIONS:
Overall Officials: Karin Tanja-Dijkstra, docter, Principal Investigator — University of Twente; Berend Koudstaal, Study Chair — Erasmus Medical Center
Locations (1):
- ErasmusMC, Rotterdam, South Holland, Netherlands